CLINICAL TRIAL: NCT05790668
Title: Motivational Refinements for Facilitating Reinforcement Schedule Thinning
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Brian D. Greer, Ph.D., BCBA-D, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro2021002237
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Decreasing Destructive Behavior; Increasing Functional Communicative Behavior
Keywords: functional communication training; reinforcement schedule thinning; resurgence; treatment relapse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Evaluation of PIA-Informed Schedule Thinning (Experimental): The goal of Arm 1 will be to will extend pilot work on the utility of individualizing the starting point for reinforcement schedule thinning based on the results of a progressive-interval assessement (PIA). The investigators will do so by conducting reinforcement schedule thinning using a multielement design in two separate contexts, one informed by the results of a PIA and another not so informed. The criteria for schedule thinning will be identical across both conditions but will be applied to each condition independently. Investigators will determine the efficiency of schedule thinning, reductions of destructive behavior, and durability of functional communication responses across the two conditions.
  Interventions: Behavioral: Traditional Schedule Thinning; Behavioral: PIA-Informed Schedule Thinning
- Evaluation of Competing Items (Experimental): The goal of Arm 2 will be to evaluate the utility of competing items (e.g., alternative reinforcement or activities) during schedule thinning. Both conditions will be informed by the PIA, similar to the experimental condition in Arm 1. PIA-informed schedule thinning with competing stimuli will be identical to that of PIA-informed schedule thinning, except (a) the therapist will provide continuous access to the highly competing stimulus identified by that participant's competing stimulus assessment (e.g., providing attention while an iPad is unavailable, playing music while working), and (b) it will occur in the other context (e.g., the yellow context). Investigators will determine the efficiency of schedule thinning, reductions of destructive behavior, the durability of functional communication responses across the two conditions, and resurgence of destructive behavior during prolonged periods of extinction.
  Interventions: Behavioral: PIA-Informed Schedule Thinning; Behavioral: PIA-Informed Schedule Thinning with Competing Stimuli
- Effects of Competing Items on PIA Outcomes (Experimental): The goal of Arm 3 will be to examine potential interaction effects between the above two experimental arms by conducting PIAs with no, low, moderate, and high competing stimuli to determine the schedule duration at which schedule thinning should commence with each competing stimulus. All participants will complete this arm prior to enrollment in Arms 1 or 2. The investigators will randomize the sequence of each of the four PIAs (PIA with no competing stimuli, PIA with low competing stimuli, PIA with moderately competing stimuli, PIA with highly competing stimuli) across participants.
  Interventions: Behavioral: PIA-Informed Schedule Thinning with Competing Stimuli

INTERVENTIONS:
Behavioral: Traditional Schedule Thinning — During traditional schedule thinning during functional communication training with discriminative stimuli (e.g., multiple schedules, chained schedules), practitioners correlate a unique stimulus with reinforcement (e.g., a green card) and another for extinction (e.g., a red card). When the reinforcement and extinction stimuli are presented, the child's communication responses are honored or not honored, respectively. Behavior analysts begin with a brief period of extinction (e.g., 2 s) and gradually increase that duration as the child displays low levels of destructive behavior and high levels of discriminated communication responses (i.e., communication requests during reinforcement components only) until the child reaches a terminal schedule informed by caregiver/child preference (e.g., 2.5-min reinforcement, 10-min extinction). Typically, the starting extinction period is brief and arbitrarily selected and there are no competing stimuli programmed.
  Arms: Evaluation of PIA-Informed Schedule Thinning
Behavioral: PIA-Informed Schedule Thinning — This intervention involves the same general components as Traditional Schedule Thinning. However, rather than starting with an arbitrary duration of the extinction component (e.g., 2 s), the behavior analyst empirically derives the starting point based on a progressive-interval assessment (PIA). The PIA involves rapidly increasing the duration of the extinction component within a single session to determine the leanest schedule of reinforcement that does not produce untoward effects. Behavior analysts will progress through the following extinction durations within a single session: 3 s, 11 s , 21 s, 34 s, 50 s, 70 s, 95 s, 126 s, 164 s, 213 s, and 270 s. For example, if the participant displays destructive behavior at 164 s consistently, but not at 126 s, the experimenters will start schedule thinning with a 126-s extinction component. There will be no competing stimuli programmed in this intervention.
  Arms: Evaluation of Competing Items; Evaluation of PIA-Informed Schedule Thinning
Behavioral: PIA-Informed Schedule Thinning with Competing Stimuli — This intervention is identical to PIA-Informed Schedule Thinning except that behavior analysts will program competing activities (e.g., alternative activities like toys or therapist attention) during extinction components. The competing stimuli will be derived from a competing stimulus assessment in which destructive behavior is analyzed across various conditions in which only the activity is manipulated during the extinction period (e.g., a session with action figures during extinction, a session with tablet during extinction). The items that produce the highest levels of child engagement and lowest levels of destructive behavior are known as highly competing items.
  Arms: Effects of Competing Items on PIA Outcomes; Evaluation of Competing Items

SUMMARY:
Destructive behavior represents a comorbid condition of developmental disability for which risk increases with intellectual disability severity, communication deficits, and co-occurring autism spectrum disorder. Destructive behavior, such as self-injurious behavior and aggression, causes harm to the child and others and increases the risk for institutionalization, social isolation, physical restraint, medication overuse, and abuse. Clinicians have used functional analyses to identify the variables that reinforce destructive behavior and to develop effective, function-based treatments. Functional communication training (FCT) is an empirically supported, function-based treatment that decreases destructive behavior. Using FCT, the clinician teaches the child to use a functional communication response (FCR) to request the reinforcer maintaining destructive behavior, while placing destructive behavior on extinction. For example, if functional analysis results showed that attention reinforced destructive behavior, the clinician would provide attention when the child used the FCR ("Play with me, please") and would not provide attention for destructive behavior. Two limitations of FCT are that (a) schedules of reinforcement maintaining the FCR must often be thinned gradually to levels that are practical for caregivers to implement consistently in the home and in the community, and (b) this necessary process of reinforcement schedule thinning regularly causes destructive behavior to increase following initially effective treatment, a form of treatment relapse called resurgence. The current project aims to improve these limitations of FCT by (a) hastening the process of reinforcement schedule thinning by removing unnecessary schedule-thinning steps using the results of a progressive interval assessment and (b) mitigating the resurgence of destructive behavior by providing stimuli that highly compete with the reinforcer maintaining destructive behavior. The investigators will conduct a randomized clinical trial to evaluate the extent to which these two promising refinements to FCT improve the process of reinforcement schedule thinning, and an exploratory experiment will examine the interactive effects of these two approaches. This novel project has the potential to substantially improve standards of care guiding the treatment of severe destructive behavior and to improve the long-term outcomes for children and families afflicted by these debilitating behavior disorders.

DETAILED DESCRIPTION:
The severe destructive behavior (e.g., self-injury, aggression) of children with intellectual developmental disorder is prevalent, often dangerous, and negatively impacts social integration and quality of life (Borthwick-Duffy, 1994; Crocker et al., 2006). Function-based interventions that rely on differential reinforcement of alternative behavior reduce such problematic behavior effectively (Greer et al., 2016; Hagopian et al., 1998; Rooker et al., 2013), but the clinical utility of this approach is hampered in two critically important ways. First, schedules of reinforcement maintaining alternative behavior must be thinned to levels that are practical for caregivers to implement consistently in the home and in the community (Greer et al., 2016; Hagopian et al., 2011). This necessary process of schedule thinning often requires substantial time and resources to complete and typically comprises the most expensive portion of routine, clinical service delivery for this referral concern. Second, and exacerbating the first, is the consistent finding that schedule thinning often produces a form of treatment relapse called resurgence (Briggs et al., 2018; Mitteer et al., 2022; Muething et al., 2020; Shahan et al., 2020). The experimenters propose two clinically indicated, and theoretically grounded, methods of accelerating the process of schedule thinning while mitigating the resurgence of severe destructive behavior.

Recent research from the investigators has shown that the quantitative theory of resurgence called Resurgence as Choice (RaC) (Greer & Shahan, 2019; Shahan et al., 2019; Shahan & Craig, 2017) accurately describes how decrements in the availability of reinforcement predict the amount of resurgence of destructive behavior during the process of schedule thinning (Shahan & Craig, 2017), a finding recently verified in a nonhuman animal study (Shahan et al., 2020). Importantly, clinical and laboratory research alike has shown, as RaC predicts, that simply thinning reinforcement in small, gradual steps, the approach most commonly used by clinicians, does not prevent resurgence-relapse inevitably occurs once the schedule reaches a break point (Briggs et al., 2018; Shahan et al., 2020; Shahan & Craig, 2017; Shahan & Greer, 2021). RaC theory states that motivation for the functional reinforcer maintaining destructive behavior (parameter a in RaC equations) plays an important role in determining whether and to what extent destructive behavior will resurge during schedule thinning (Greer et al., 2019; Shahan et al., 2019; Shahan & Craig, 2017), a prediction well-supported by recent pilot work from the investigators on (a) individualizing the starting point for schedule thinning using a progressive interval assessment (PIA) (Miller et al., 2021) and (b) providing competing stimuli to hasten schedule thinning (Fuhrman et al, 2018; Miller et al., 2021). According to RaC theory, these two clinically indicated manipulations facilitate schedule thinning by respectively (a) tailoring the initial schedule of reinforcement to each patient's unique level of motivation for the functional reinforcer and (b) dampening motivation for the functional reinforcer by delivering an alternative and competing source of reinforcement. Additionally, theoretical and empirical work in the area of behavioral economics provides independent support for these two manipulations. This project will further the clinical and theoretical understanding of how motivational variables affect resurgence as it occurs in practice, and the project has the potential to substantially improve standards of care guiding the treatment of severe destructive behavior.

The experimenters will conduct a study to identify whether quantitatively informed refinements can improve efficiency and efficacy of reinforcement schedule thinning when treating severe destructive behavior. The project has three specific aims:

Specific Aim 1: The experimenters will extend pilot work on the utility of individualizing the starting point for reinforcement schedule thinning based on the results of a PIA. The experimenters will accomplish this by conducting reinforcement schedule thinning in two distinct stimulus contexts, one informed by the results of a PIA and another not so informed.

Specific Aim 2: Basing the starting point on a PIA, the experimenters will assess the extent to which providing competing stimuli from a competing stimulus assessment quickens the process of schedule thinning when competing stimuli are available in one, but not another, unique stimulus context.

Specific Aim 3: The experimenters will examine the potential interaction effects between these two approaches by conducting PIAs with no, low, moderate, and high competing stimuli to determine the schedule duration at which schedule thinning should commence with each competing stimulus.

ELIGIBILITY:
Inclusion Criteria:

* boys and girls from ages 3 to 17
* destructive behavior that occurs at least 10 times a day, despite previous treatment
* destructive behavior reinforced by social consequences
* stable protective supports for self-injurious behavior (e.g., helmet) with no anticipated changes during enrollment
* on a stable psychoactive drug regimen for at least 10 half-lives per drug or drug free
* stable educational plan and placement with no anticipated changes during the child's treatment

Exclusion Criteria:

* patients who do not meet the inclusion criteria
* patients currently receiving 15 or more hours per week of treatment for their destructive behavior
* Diagnostic and Statistical Manual-5 diagnosis of Rett syndrome or other degenerative conditions (e.g., inborn error of metabolism)
* a comorbid health condition or major mental disorder that would interfere with study participation
* occurrence of self-injury during study assessments that presents a risk of serious or permanent harm (e.g., detached retinas) based on routine clinical-risk assessment
* patients requiring changes to protective supports for self-injury or drug treatment, but investigators will invite these patients to participate when protective supports and drug regimen are stable

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Destructive behavior (responses per minute) | Through study completion, an average of 4 weeks.
  The primary outcome measure is responses per minute of destructive behavior. The investigators will calculate this outcome by dividing the total number of destructive responses per session by the total number of minutes spent in session.
Discriminated functional communication responses (percentage) | Through study completion, an average of 4 weeks.
  The investigators will calculate this outcome by dividing the number of child requests when reinforcement is signaled as available by the total number of child requests during reinforcement and extinction, then multiplying the quotient by 100 to convert it to a percentage. This indicates the level of accuracy with communication requests, with 80-100% being optimal.
Efficiency of schedule thinning | Through study completion, an average of 4 weeks.
  In addition to the above metrics, it is expect that informing schedule thinning with the PIA or competing items may result in reaching the terminal schedule (e.g., 270-s extinction) more rapidly than conditions not so informed. Thus, investigators will analyze the number of treatment sessions required for an intervention to produce destructive behavior below an 85% reduction from baseline and discriminated functional communication responses above 80% at the terminal-schedule value.

CONTACTS AND LOCATIONS:
Overall Officials: Brian D Greer, Ph.D., Principal Investigator — Rutgers, The State University of New Jersey
Locations (2):
- United States (2):
  - Douglass Developmental Disabilities Center, New Brunswick, New Jersey
  - Rutgers University Center for Autism Research, Education, and Services, Somerset, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share outcome data using the National Database on Autism Research (NDAR). The investigators will also share outcome data on the human participants in these two experiments who are not diagnosed with autism spectrum disorder to better understand how complex, comorbid disorders (e.g., self-injury) differ in individuals with and without autism spectrum disorder.
Supporting Information: Study Protocol, SAP
Time Frame: Within one year of the primary completion date of the studies.
Access Criteria: In accordance with NDAR policy.

REFERENCES:
- [Background] Borthwick-Duffy SA. Epidemiology and prevalence of psychopathology in people with mental retardation. J Consult Clin Psychol. 1994 Feb;62(1):17-27. doi: 10.1037//0022-006x.62.1.17. PMID 8034819
- [Background] Briggs AM, Fisher WW, Greer BD, Kimball RT. Prevalence of resurgence of destructive behavior when thinning reinforcement schedules during functional communication training. J Appl Behav Anal. 2018 Jul;51(3):620-633. doi: 10.1002/jaba.472. Epub 2018 May 17. PMID 29774545
- [Background] Crocker AG, Mercier C, Lachapelle Y, Brunet A, Morin D, Roy ME. Prevalence and types of aggressive behaviour among adults with intellectual disabilities. J Intellect Disabil Res. 2006 Sep;50(Pt 9):652-61. doi: 10.1111/j.1365-2788.2006.00815.x. PMID 16901292
- [Background] Fuhrman AM, Greer BD, Zangrillo AN, Fisher WW. Evaluating competing activities to enhance functional communication training during reinforcement schedule thinning. J Appl Behav Anal. 2018 Oct;51(4):931-942. doi: 10.1002/jaba.486. Epub 2018 Jun 29. PMID 29959773
- [Background] Greer BD, Fisher WW, Saini V, Owen TM, Jones JK. Functional communication training during reinforcement schedule thinning: An analysis of 25 applications. J Appl Behav Anal. 2016 Mar;49(1):105-21. doi: 10.1002/jaba.265. Epub 2015 Oct 20. PMID 26482103
- [Background] Greer BD, Shahan TA. Resurgence as Choice: Implications for promoting durable behavior change. J Appl Behav Anal. 2019 Jul;52(3):816-846. doi: 10.1002/jaba.573. Epub 2019 May 3. PMID 31049954
- [Background] Hagopian LP, Boelter EW, Jarmolowicz DP. Reinforcement schedule thinning following functional communication training: review and recommendations. Behav Anal Pract. 2011 Summer;4(1):4-16. doi: 10.1007/BF03391770. PMID 22532899
- [Background] Hagopian LP, Fisher WW, Sullivan MT, Acquisto J, LeBlanc LA. Effectiveness of functional communication training with and without extinction and punishment: a summary of 21 inpatient cases. J Appl Behav Anal. 1998 Summer;31(2):211-35. doi: 10.1901/jaba.1998.31-211. PMID 9652101
- [Background] Miller SA, Fisher WW, Greer BD, Saini V, Keevy MD. Procedures for determining and then modifying the extinction component of multiple schedules for destructive behavior. J Appl Behav Anal. 2022 Mar;55(2):463-480. doi: 10.1002/jaba.896. Epub 2021 Dec 12. PMID 34897677
- [Background] Mitteer DR, Greer BD, Randall KR, Haney SD. On the scope and characteristics of relapse when treating severe destructive behavior. J Appl Behav Anal. 2022 Jun;55(3):688-703. doi: 10.1002/jaba.912. Epub 2022 Mar 15. PMID 35290666
- [Background] Muething C, Pavlov A, Call N, Ringdahl J, Gillespie S. Prevalence of resurgence during thinning of multiple schedules of reinforcement following functional communication training. J Appl Behav Anal. 2021 Apr;54(2):813-823. doi: 10.1002/jaba.791. Epub 2020 Oct 25. PMID 33103244
- [Background] Rooker GW, Jessel J, Kurtz PF, Hagopian LP. Functional communication training with and without alternative reinforcement and punishment: an analysis of 58 applications. J Appl Behav Anal. 2013 Dec;46(4):708-22. doi: 10.1002/jaba.76. Epub 2013 Aug 22. PMID 24114463
- [Background] Shahan TA, Browning KO, Nall RW. Resurgence as Choice in Context: Treatment duration and on/off alternative reinforcement. J Exp Anal Behav. 2020 Jan;113(1):57-76. doi: 10.1002/jeab.563. Epub 2019 Nov 27. PMID 31777091
- [Background] Shahan TA, Browning KO, Nist AN, Sutton GM. Resurgence and downshifts in alternative reinforcement rate. J Exp Anal Behav. 2020 Sep;114(2):163-178. doi: 10.1002/jeab.625. Epub 2020 Aug 27. PMID 32856313
- [Background] Shahan TA, Craig AR. Resurgence as Choice. Behav Processes. 2017 Aug;141(Pt 1):100-127. doi: 10.1016/j.beproc.2016.10.006. Epub 2016 Oct 26. PMID 27794452
- [Background] Shahan TA, Greer BD. Destructive behavior increases as a function of reductions in alternative reinforcement during schedule thinning: A retrospective quantitative analysis. J Exp Anal Behav. 2021 Sep;116(2):243-248. doi: 10.1002/jeab.708. Epub 2021 Jul 4. PMID 34219242